CLINICAL TRIAL: NCT04113629
Title: Evaluation of Simplified HCV Diagnostics in HIV/HCV Co-infected Patients in Myanmar (Simplified Monitoring Myanmar SM2 Study)
Brief Title: Simplified Monitoring Myanmar SM2 Study
Acronym: SM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: University of Public Health, Myanmar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VHCRP1803
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C; Liver Cirrhoses; Liver Inflammation; HIV Infections
MeSH Terms: conditions — Hepatitis C; Hepatitis; HIV Infections

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sofosbuvir/Daclatasvir (Other): standard DAA therapy: 12 or 24 weeks of sofosbuvir/daclatasvir
  Interventions: Device: HCV point of care machine

INTERVENTIONS:
Device: HCV point of care machine — Xpert HCV Assay performed on the GeneXpert point of care machine

SUMMARY:
The study will evaluate the proportion of patients with undetectable HCV RNA at 12 weeks post-treatment (SVR12) following a course of DAA therapy delivered using a simplified schedule of safety and virological monitoring.

DETAILED DESCRIPTION:
A total of 200 HIV/HCV co-infected patients who plan to commence DAA therapy at Specialist Hospital Waibargi and Mingaladon, will be enrolled by simple random sampling.

In addition to standard of care medical procedures, each participant will complete a questionnaire and have blood taken for standard HCV RNA testing.

They will also have a finger-stick capillary blood sample collected for a HCV point of care test, using the the Xpert HCV Assay performed in the GeneXpert point of care machine.

Dried blood spot collection (DBS) for HCV core antigen and HCV RNA testing will be collected as a research sample. Concordance between standard of care method and new DBS method will be evaluated.

The proportion of patients reaching SVR will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to participate in this study.

1. Have voluntarily signed the consent form.
2. 18 years of age or older.
3. HCV antibody positive.
4. HIV antibody positive.

Exclusion Criteria:

Subjects who meet any of the exclusion criteria are not to be enrolled in this study.

1. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with the subject treatment, assessment or compliance with the protocol.
2. Creatinine clearance (CLcr) < 30mL/min at screening.
3. Pregnant or nursing female.
4. Use of prohibited concomitant medications.
5. Inability or unwillingness to provide informed consent or abide by the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with undetectable HCV RNA at 12 weeks post-treatment (SVR12) | 12 weeks post completion of commenced treatment
  To evaluate the proportion of patients with undetectable HCV RNA at 12 weeks post-treatment (SVR12) following a course of DAA therapy delivered using a simplified schedule of safety and virological monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- The Kirby Institute, University of New South Wales Australia, Sydney, New South Wales, Australia